CLINICAL TRIAL: NCT03677713
Title: Nasal Packing Following Endoscopic Endonasal Pituitary Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Principal Investigator, Shaun Kilty, MD, FRCSC, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20180541-01H
Record Dates: First submitted 2018-07-06; First posted 2018-09-19 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Pituitary Tumor
Keywords: endoscopic; endonasal; transsphenoidal; surgical resection; pituitary tumour; nasal packing; Merocel
MeSH Terms: conditions — Pituitary Neoplasms

STUDY DESIGN:
Intervention Model Description: A single center, non-blinded, randomized controlled trial (RCT) will be conducted as a pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nasal Packing (Active Comparator): Nasal packing will be placed at the end of surgery.
  Interventions: Procedure: Nasal Packing
- No Nasal Packing (Experimental): No nasal packing will be placed during or after the surgery.
  Interventions: Procedure: No nasal packing.

INTERVENTIONS:
Procedure: No nasal packing. — No nasal packing at the end of the surgery
  Arms: No Nasal Packing
Procedure: Nasal Packing — Patients will have nasal packing at the end of the surgery
  Arms: Nasal Packing

SUMMARY:
There is considerable controversy about the use of nasal packing following endoscopic endonasal resection of pituitary tumors as a necessary treatment amongst Rhinology-Skull Base Surgeons. The justification for the routine use of nasal packing following pituitary surgery is not clear as this practice is not used for equally extensive sinus surgery. Further scientific evidence supporting this practice is lacking, and a recent survey of Canadian surgeons performing this surgery demonstrates clear division in practice for the routine use of nasal packing. Nasal packing causes patients significant discomfort requiring medication, and the use of packing adds direct and unintended hospitalization and health system costs for every case for which it is used. The benefits, short-comings, and associated costs of nasal packing following endoscopic endonasal transsphenoidal pituitary resection have not been studied.

OBJECTIVE: To determine if nasal packing following endoscopic endonasal pituitary tumor surgery is a necessary treatment. The principal research questions for this study, our internal pilot of the RCT, pertain to feasibility of enrolment of patients undergoing endoscopic endonasal transsphenoidal pituitary tumor surgery using the full RCT protocol of nasal packing versus no nasal packing. The pilot will address feasibility of site-specific enrolment and feasibility of institutional ethics approval and protocol administration.

DETAILED DESCRIPTION:
BACKGROUND AND CLINICAL SIGNIFICANCE

Over the past decade, the surgical method for removing pituitary tumors has shifted from a microscopic resection technique performed exclusively by a neurosurgeon, to an endoscopic resection done as a team with an otolaryngologist and neurosurgeon. This field continues to evolve given this recent shift in treatment technique.

Nasal packing has historically been a post-operative intervention of treating the nose employed by otolaryngologists for any nasal surgery they performed. However, with the advent of endoscopic sinus surgery and changes in surgical technique, the use of nasal packing has become less common. A systematic review by Quinn et. Al (2013) showed that nasal packing caused more patient discomfort than any other post-septoplasty maneuver and did not prevent complications of septoplasty, but could contribute to adverse events following septoplasty. In North America, nasal packing is no longer commonly used after septoplasty.

However, following the endoscopic resection of pituitary tumors, the practice of nasal packing is still widely employed. The reasoning for placement of nasal packing following surgery is not clear, just as it was not for its use following septoplasty. A thorough search of the literature did not identify any publications providing justification for the use of nasal packing. Published recommendations to reduce incidence of post-operative nasal complications after transsphenoidal pituitary tumor resection include use of specific nasal medications (intranasal corticosteroids) and regular nasal saline irrigation (in patients without cerebrospinal fluid rhinorrhea) to clear nasal mucosal hyperemia edema and secretions, as well as to prevent nasal synechiae and scarring, to maintain the sinus cavity drainage, and accelerate the recovery of the physiological function of the paranasal sinus. However, an evidence based recommendation in support or against routine nasal packing has not been made. A review from neurosurgical literature on perioperative management post transsphenoidal pituitary resection reports the majority of patients do not require insertion of nasal packing at the time of surgery, some patients (intraoperative Cerebral spinal fluid (CSF) leaks requiring sellar floor reconstruction, Cushing's Disease, and acromegaly) may benefit from their insertion, and if used packing is typically removed postoperative day 1.

In January 2018 an informal email survey of Canadian Otolaryngologists who routinely perform endoscopic pituitary surgery with a neurosurgeon (total of 7 respondents out of 11 surgeons, 64% response rate) demonstrated that 5 of 7 use nasal packing following the procedure; 2 of 7 do not. Packing is usually left in place for 48 hours when used. A screening of institution websites (February 12, 2018) in North America where this surgery is routinely performed found a balanced number of institutions that list the use or non-use of nasal packing following endoscopic pituitary tumor resection (13 institutional websites screened, 8 institutions routinely use nasal packing, 5 do not). There is clinical equipoise related to the use of nasal packing. An objective study assessing the utility of nasal packing following endoscopic endonasal pituitary surgery has not yet been completed.

This study seeks to answer the question, "Is routine nasal packing following endoscopic pituitary tumor surgery a necessary treatment?". The results of this trial have the potential to standardize practice patterns in Canada and internationally, and will inform evidence based practice while directly impacting the quality of care delivered to patients undergoing pituitary tumor resection.

HYPOTHESIS

Nasal packing following routine endoscopic pituitary tumor surgery is an unnecessary intervention that may cause patients unjustified post-operative discomfort, negatively affect their quality of life, and unnecessarily increase associated cost of care.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* undergoing endoscopic endonasal transsphenoidal approach to pituitary resection for pituitary tumors of any pathology for the first time

Exclusion Criteria:

* patients who do not have a working understanding of English
* patients with known allergy to Merocel nasal packing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Anterior Skull Basal Nasal Inventory-12 (ASK-12) | Post Op Day 0, 1, 2, 3 and Post-Op weeks 2 and 4
  The ASK-12 is a validated patient reported nasal QOL questionnaire that evaluates morbidity after endonasal skull base surgery. Twelve symptoms related to nasal health are scored 0-5 and a global score is the mean value. Lower scores reflect better sinonasal quality of life.
Incidence of sinonasal adverse events | Post Op Day 0, 1, 2, 3 and Post-Op weeks 2 and 4
  Evaluated by comparing the proportion of patients in each group who develop any sinonasal adverse events ( epistaxis, sinusitis, synechia, CSF rhinorrhea, nasal septal perforation

SECONDARY OUTCOMES:
Change in EuroQual-5Dimension (EQ-5D) | Post Op Day 0, 1, 2, 3 and Post-Op weeks 2 and 4
  Quality of Life Survey
Cost Analysis | Through study completion, 1 year.
  An analysis of the direct and indirect costs related to hospitalization and medication use.
Change in Analgesic and Antibiotic Usage | Post Op Day 0, 1, 2, 3 and Post-Op weeks 2 and 4
  The total amount (dosage) of analgesic and antibiotics administered during the study period.
Post operative pain | Post Op Day 0, 1, 2, 3 and Post-Op weeks 2 and 4
  Will be captured using a visual analogue scale (VAS). Scores range from 0 to 10. Lower score indicate less severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Shaun Kilty, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No